CLINICAL TRIAL: NCT07119801
Title: Clinical and Ultrasonographic Evaluation of the Efficacy of Extracorporeal Shock Wave Therapy (ESWT) in Post-Stroke Spasticity: A Randomized Controlled Trial
Brief Title: Clinical and Ultrasonographic Evaluation of the Efficacy of Extracorporeal Shock Wave Therapy (ESWT) in Post-Stroke Spasticity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Meltem Gunes Akinci, Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleU.ftr-MGAkıncı-001
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Spastic Hemiplegia; Extracorporal Shockwave Therapy (ESWT)
Keywords: spastic hemiplegia; extracorporeal shockwave therapy; spasticity of the wrist flexors
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): This group will receive physical therapy for 1-2 hours daily, 5 days a week, for 12 weeks. The therapy will include range of motion (ROM) exercises, stretching exercises, progressive resistive exercises, positioning, postural control, weight-bearing exercises, balance and gait training, and occupational therapy. Speech and language therapy will also be included according to the patient's needs.
  Interventions: Other: Conventional rehabilitation
- radial ESWT (rESWT) plus conventional rehabilitation group (Experimental): The rESWT will be applied to the Flexor Carpi Ulnaris (FCU) and Flexor Carpi Radialis (FCR) muscles twice a week for four weeks, totaling eight sessions. The application site will be the midpoint of the most prominent part of each muscle. For each muscle, a 15 mm applicator head will be used to deliver 2000 impulses at a frequency of 5 Hz and an intensity of 60 mJ (1 bar), corresponding to an energy flux density of 0.340 mJ/mm². Additionally, this group will receive physical therapy for 1-2 hours daily, 5 days a week, for 12 weeks. The therapy will include range of motion (ROM) exercises, stretching exercises, progressive resistive exercises, positioning, postural control, weight-bearing exercises, balance and gait training, and occupational therapy. Speech and language therapy will also be included according to the patient's needs.
  Interventions: Device: Radial Extracorporeal Shock Wave Therapy; Other: Conventional rehabilitation

INTERVENTIONS:
Device: Radial Extracorporeal Shock Wave Therapy — rESWT will be administered to the FCU and FCR muscles two days per week over a period of four weeks (8 sessions in total). The point of application will be selected as the center of the muscle belly for both the FCU and FCR. Each muscle will receive 2000 shocks using a 15 mm applicator tip at a frequency of 5 Hz. The treatment will be conducted at an intensity of 60 mJ (1 bar), with an energy flux density of 0.340 mJ/mm².
  Arms: radial ESWT (rESWT) plus conventional rehabilitation group
Other: Conventional rehabilitation — Conventional rehabilitation will be administered for 1-2 hours daily, 5 days a week, for 12 weeks. It will include range of motion exercises, stretching exercises, progressive resistive exercises, positioning, postural control, weight shifting, balance, gait training, occupational therapy, and speech-language therapy according to the patient's needs.

SUMMARY:
This research evaluate the effectiveness of Extracorporeal Shock Wave Therapy (ESWT) for treating spasticity in the wrist flexor muscles (flexor carpi ulnaris - FCU and flexor carpi radialis - FCR) of chronic stroke patients.

Spasticity, a common complication after a stroke, causes muscle stiffness, pain, and functional limitation, leading to increased healthcare costs and a lower quality of life. Current treatments like medication and injections have significant drawbacks, such as side effects and high costs, creating a need for new, non-invasive, and effective methods.

The study highlights that traditional methods for assessing spasticity, like the Modified Ashworth Scale (MAS), are subjective. It proposes using objective, non-invasive ultrasound techniques-specifically strain elastography (to measure muscle stiffness) and echogenicity (to assess muscle tissue quality)-for a more reliable evaluation.

The primary goal of this research is to be the first to investigate the short- and long-term effects of ESWT on the FCR and FCU muscles using these objective ultrasound measures alongside traditional clinical scales. The findings are expected to help standardize ESWT treatment protocols and promote the use of objective ultrasound data for the management and follow-up of post-stroke spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 65 years.
* First-ever stroke episode confirmed by MRI and/or CT scan.
* Clinical diagnosis of hemiplegia.
* More than 6 months post-stroke.
* A Modified Ashworth Scale (MAS) score between 1 and 3 for wrist flexor spasticity.

Exclusion Criteria:

* History of more than one stroke episode
* Stroke onset more than ten years ago
* Stroke onset less than 6 months ago
* Age over 65 (to limit the effects of aging on muscle structure)
* Contraindications for ESWT (e.g., cancer, local tumor or active infection in the treatment area, pregnancy, coagulation disorders, pacemaker or other electronic/metallic implants)
* Severe aphasia or serious communication problems
* Presence of fixed contracture in the wrist
* Patients who have received botulinum toxin or phenol nerve block injections within the last 6 months
* Medically unstable patients (e.g., uncontrolled hypertension, diabetes mellitus, or severe cardiac, hepatic, or renal disease)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | Baseline, 4th week, 8th week and 12th week after treatment.
  The Ashworth Scale assesses the resistance encountered when an evaluator moves a limb through its full range of motion.
  According to the Modified Ashworth Scale:
  0: No increase in muscle tone.
  1: Slight increase in muscle tone, characterized by a catch and release or by minimal resistance at the end of the range of motion.
  1+: Slight increase in muscle tone, characterized by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion.
  2: More marked increase in muscle tone throughout most of the range of motion, but the affected part(s) can be moved easily.
  3: Considerable increase in muscle tone; passive movement is difficult.
  4: Affected part(s) are rigid in flexion or extension.

SECONDARY OUTCOMES:
Wrist range of motion | Baseline 4th week 8th week and 12th week after treatment.
  During the measurement, the goniometer is aligned with the joint's axis of rotation to determine the maximum angle during passive movement. It is crucial that the limb is moved slowly and carefully to avoid eliciting resistance from the patient's spastic muscles. A slow, controlled movement minimizes spasticity, thereby ensuring a more accurate measurement.Wrist passive range of motion will be measured.
Modified Barthel Index | Baseline, 4th week, 8th week and 12th week after treatment.
  The Barthel Index (BI) consists of 10 items related to mobility and activities of daily living (ADL), and it assesses activities such as feeding, transfer from wheelchair to bed and back, personal grooming, bathing, walking, ascending and descending stairs, dressing, and bladder and bowel continence.
  The Modified Barthel Index (MBI) is a revision of the original Barthel Index (BI) and uses the same 10 items. The main difference between these two measures is that the MBI consistently classifies patient performance into five scoring levels: unable to perform the task, attempts the task but is unsafe, moderate assistance required, minimal assistance required, and fully independent. The total score of the MBI also ranges from 0 to 100, with higher scores indicating greater independence in ADL.
The Fugl-Meyer Upper Extremity Scale | Baseline, 4th week, 8th week and 12th week after treatment.
  The Fugl-Meyer Assessment for the Upper Extremity (FMA-UE) is designed to quantitatively evaluate the motor function of stroke patients and includes tests for upper extremity motor and sensory function. The FMA-UE is used to assess upper extremity motor impairment and contains 33 items scored on a scale from 0 to 2 (0 = cannot perform, 1 = performs partially, and 2 = performs fully), with a total score range of 0-66. The FMA has been reported to have high reliability for testing motor performance in post-stroke patients.
Modified Heckmatt Scale | Baseline, 4th week, 8th week and 12th week after treatment.
  he Modified Heckmatt Scale is a method that uses ultrasonography to reliably evaluate echogenic changes in a spastic muscle, thereby indicating the level of fibrotic change. The Modified Heckmatt Scale was developed to achieve greater sensitivity between grades compared to the original Heckmatt Scale, particularly for muscles with mildly to moderately increased echo intensity (Grades 2 and 3).
  Grade 1: Normal echogenicity, distinct from the bone echo, is observed in over 90% of the muscle.
  Grade 2: There is increased muscle echogenicity in 10-50% of the tissue, but a distinct bone echo and areas of normal muscle echo are still present.
  Grade 3: A marked increase in muscle echogenicity is seen in 50% to 90% of the tissue, with reduced differentiation of the bone echo from the muscle.
  Grade 4: Very strong muscle echogenicity is observed in >90% of the tissue, with a near-complete loss of the distinct bone echo from the muscle.
Sonoelastographic strain index | Baseline, 4th week, 8th week and 12th week after treatment.
  Quantitative elastography analysis will be used to measure stiffness. As a software feature of the ultrasound system, quantitative elastography analysis numerically measures the color distribution in a selected area across single or multiple frames and calculates an elasticity index for the measured area.
  The elasticity index is a value between 0.0 and 6.0, generated by the reflected color distribution within the selected region. A higher value signifies greater stiffness, which is predominantly represented by the color blue on the screen. While the elasticity index is calculated separately for the reference area and the muscle, the system automatically calculates the strain ratio as muscle/reference area.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Güneş Akıncı, Assistant professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)